CLINICAL TRIAL: NCT03498352
Title: Rest Ventilatory Parameters Predict Morbidity and Mortality in Patients Undergoing Thoracic Surgery
Brief Title: Rest Ventilatory Parameters Predict Morbidity and Mortality in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Ivan Cundrle, M.D., Ph.D., St. Anne's University Hospital Brno, Czech Republic
Other Study IDs: IIT/2017/12 and 2018/08
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Complication; Cardiovascular Complication
Keywords: cardiopulmonary exercise testing, thoracic surgery
MeSH Terms: interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thoracic surgery — Lung resection surgery

SUMMARY:
Cardiopulmonary exercise testing is recommended for preoperative evaluation and risk stratification of lung resection candidates. Ventilatory efficiency (VE/VCO2 slope) has been shown to predict morbidity and mortality in lung resection candidates and has been shown superior to peak oxygen consumption (VO2). Patients with increased VE/VCO2 during exercise also exhibit increased VE/VCO2 ratio and decreased end-tidal CO2 at rest. Our first hypothesis is that rest ventilatory parameters predict morbidity and mortality in patients undergoing thoracic surgery. VE/VCO2 is well correlated with ventilation-perfusion mismatch, therefore it may be useful in hypoxemia prediction during one-lung ventilation during thoracic surgery. Our second hypothesis is that patients with high VE/VCO2 will be prone to hypoxemia development during one-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* thoracotomy because of lung infiltration (confirmed or highly suspicious lung tumor)

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients planned for thoracotomy because of lung infiltration (confirmed or highly suspicious lung tumor). Patients will be recruited from 2 centers in the Czech Republic (St. Anne's University Hospital, Brno, Czech Republic and University Hospital in Brno).
Sampling Method: Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary complications | Respiratory complications will be assessed from the first 30 post-operative days or from the hospital stay.
  Respiratory complications definition: pneumonia, atelectasis; respiratory failure needing mechanical ventilation; adult respiratory distress syndrome; pneumothorax present on the 3rd post-operative day; long-lasting pleural effusions present on the 3rd post-operative day

SECONDARY OUTCOMES:
Intensive care length of stay | From the first 30 post-operative days or from the hospital stay.
  In all subjects, intensive care unit length of stay will be assessed.
Hospital length of stay | From the first 30 post-operative days or from the hospital stay.
  In all subjects, hospital length of stay will be assessed.
Cardiovascular complications | Cardiovascular complications will be assessed from the first 30 post-operative days or from the hospital stay.
  Cardiovascular complications definition: new arrhythmias (atrial fibrillation, supraventricular tachycardia, etc.); hypotension; heart failure; pulmonary edema; pulmonary embolism; myocardial infarction/minimal myocardial lesion; cardiopulmonary resuscitation
Mortality | 30 and 90 days after surgery.
  In all subjects, 30 and 90 days mortality will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cundrle, M.D., Ph.D., Principal Investigator — St. Anne's University Hospital Brno
Locations (2):
- Czechia (2):
  - University Hospital Brno, Brno, Czech Republic
  - St. Anne's University Hospital Brno, Brno, Czech Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunelli A, Belardinelli R, Pompili C, Xiume F, Refai M, Salati M, Sabbatini A. Minute ventilation-to-carbon dioxide output (VE/VCO2) slope is the strongest predictor of respiratory complications and death after pulmonary resection. Ann Thorac Surg. 2012 Jun;93(6):1802-6. doi: 10.1016/j.athoracsur.2012.03.022. Epub 2012 May 4. PMID 22560968
- [Background] Choi H, Mazzone P. Preoperative evaluation of the patient with lung cancer being considered for lung resection. Curr Opin Anaesthesiol. 2015 Feb;28(1):18-25. doi: 10.1097/ACO.0000000000000149. PMID 25486485
- [Background] Brunelli A, Charloux A, Bolliger CT, Rocco G, Sculier JP, Varela G, Licker M, Ferguson MK, Faivre-Finn C, Huber RM, Clini EM, Win T, De Ruysscher D, Goldman L; European Respiratory Society and European Society of Thoracic Surgeons joint task force on fitness for radical therapy. ERS/ESTS clinical guidelines on fitness for radical therapy in lung cancer patients (surgery and chemo-radiotherapy). Eur Respir J. 2009 Jul;34(1):17-41. doi: 10.1183/09031936.00184308. PMID 19567600
- [Background] Arena R, Myers J, Aslam SS, Varughese EB, Peberdy MA. Peak VO2 and VE/VCO2 slope in patients with heart failure: a prognostic comparison. Am Heart J. 2004 Feb;147(2):354-60. doi: 10.1016/j.ahj.2003.07.014. PMID 14760336
- [Background] Cundrle I Jr, Johnson BD, Rea RF, Scott CG, Somers VK, Olson LJ. Modulation of ventilatory reflex control by cardiac resynchronization therapy. J Card Fail. 2015 May;21(5):367-373. doi: 10.1016/j.cardfail.2014.12.013. Epub 2015 Jan 8. PMID 25576681
- [Background] Cundrle I Jr, Somers VK, Johnson BD, Scott CG, Olson LJ. Exercise end-tidal CO2 predicts central sleep apnea in patients with heart failure. Chest. 2015 Jun;147(6):1566-1573. doi: 10.1378/chest.14-2114. PMID 25742609
- [Background] Guenoun T, Journois D, Silleran-Chassany J, Frappier J, D'attellis N, Salem A, Safran D. Prediction of arterial oxygen tension during one-lung ventilation: analysis of preoperative and intraoperative variables. J Cardiothorac Vasc Anesth. 2002 Apr;16(2):199-203. doi: 10.1053/jcan.2002.31067. PMID 11957171
- [Background] Hurford WE, Alfille PH. A quality improvement study of the placement and complications of double-lumen endobronchial tubes. J Cardiothorac Vasc Anesth. 1993 Oct;7(5):517-20. doi: 10.1016/1053-0770(93)90305-5. PMID 8268428
- [Background] Schwarzkopf K, Klein U, Schreiber T, Preussetaler NP, Bloos F, Helfritsch H, Sauer F, Karzai W. Oxygenation during one-lung ventilation: the effects of inhaled nitric oxide and increasing levels of inspired fraction of oxygen. Anesth Analg. 2001 Apr;92(4):842-7. doi: 10.1097/00000539-200104000-00009. PMID 11273912
- [Background] Slinger P, Suissa S, Triolet W. Predicting arterial oxygenation during one-lung anaesthesia. Can J Anaesth. 1992 Dec;39(10):1030-5. doi: 10.1007/BF03008370. PMID 1464128
- [Background] Slinger P, Triolet W, Wilson J. Improving arterial oxygenation during one-lung ventilation. Anesthesiology. 1988 Feb;68(2):291-5. doi: 10.1097/00000542-198802000-00022. No abstract available. PMID 3277487
- [Background] Katz Y, Zisman E, Isserles SA, Rozenberg B. Left, but not right, one-lung ventilation causes hypoxemia during endoscopic transthoracic sympathectomy. J Cardiothorac Vasc Anesth. 1996 Feb;10(2):207-9. doi: 10.1016/s1053-0770(96)80238-2. PMID 8850398
- [Background] Yokota K, Toriumi T, Sari A, Endou S, Mihira M. Auto-positive end-expiratory pressure during one-lung ventilation using a double-lumen endobronchial tube. Anesth Analg. 1996 May;82(5):1007-10. doi: 10.1097/00000539-199605000-00021. PMID 8610857
- [Background] Karzai W, Schwarzkopf K. Hypoxemia during one-lung ventilation: prediction, prevention, and treatment. Anesthesiology. 2009 Jun;110(6):1402-11. doi: 10.1097/ALN.0b013e31819fb15d. PMID 19417615
- [Background] Nomoto Y. Preoperative pulmonary blood flow and one-lung anaesthesia. Can J Anaesth. 1987 Sep;34(5):447-9. doi: 10.1007/BF03014346. PMID 3664910
- [Background] Woods PR, Olson TP, Frantz RP, Johnson BD. Causes of breathing inefficiency during exercise in heart failure. J Card Fail. 2010 Oct;16(10):835-42. doi: 10.1016/j.cardfail.2010.05.003. Epub 2010 Jun 16. PMID 20932466
- [Derived] Filakovszky A, Brat K, Tschoellitsch T, Bartos S, Mazur A, Meier J, Olson L, Cundrle I. Cardiopulmonary exercise testing before lung resection surgery: still indicated? Evaluating predictive utility using machine learning. Thorax. 2025 Oct 2:thorax-2024-221485. doi: 10.1136/thorax-2024-221485. Online ahead of print. PMID 41043965
- [Derived] Brat K, Chobola M, Homolka P, Heroutova M, Benej M, Mitas L, Olson LJ, Cundrle I. Poor ventilatory efficiency during exercise may predict prolonged air leak after pulmonary lobectomy. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):269-272. doi: 10.1093/icvts/ivz255. PMID 31630177